CLINICAL TRIAL: NCT00079469
Title: Contingency Management to Enhance Smoking Cessation for Cancer Survivors: A Proof of Concept Trial
Brief Title: Bupropion and Counseling With or Without Contingency Management to Enhance Smoking Cessation in Treating Cancer Survivors Who Continue to Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 999903308; 03-C-N308; CDR0000356037
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Cancer Survivor; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cancer survivor; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bupropion

INTERVENTIONS:
Behavioral: smoking cessation intervention
Drug: bupropion hydrochloride

SUMMARY:
RATIONALE: Contingency management is a behavioral treatment approach that provides immediate rewards for positive change in behavior such as quitting smoking. In this protocol, contingency management will be in the form of a cash reward. A smoking cessation (stop-smoking) program that combines contingency management with bupropion and counseling may be effective in helping cancer survivors stop smoking.

PURPOSE: Randomized clinical trial to compare the effectiveness of bupropion and counseling with or without contingency management in helping cancer survivors stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the feasibility of a multi-component smoking cessation intervention comprising bupropion and counseling with or without contingency management (cash reward) for cancer survivors who continue to smoke.
* Compare 7-day point-prevalence abstinence rates in patients treated with these smoking cessation interventions.

Secondary

* Determine the characteristics of these patients that predict success at quitting smoking.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 smoking cessation intervention arms.

* Arm I: Patients receive oral bupropion twice daily on weeks 1-12 and brief practical counseling (i.e., problem-solving strategies, stimulus control, stress management, and social support) on weeks 1-6.
* Arm II: Patients receive treatment as in arm I and contingency management (i.e., monetary reinforcement for not smoking) on weeks 1-6.

In both arms, treatment continues in the absence of unacceptable toxicity.

Patients are followed at 12 and 24 weeks after the completion of the smoking cessation interventions.

PROJECTED ACCRUAL: A total of 100 patients (50 per intervention arm) will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer at least 6 months before study entry

  * No carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, or CNS tumor
* Smoking history of at least 2 years

  * Smoked cigarettes daily for the past 30 days
* Completed prior cancer treatment at least 6 months, but no more than 5 years before study entry

  * Concurrent tamoxifen allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000 - 450,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 2 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine < 2.0 mg/dL

Cardiovascular

* No unstable cardiovascular disease, including any of the following:

  * High-grade atrioventricular block
  * Neurocardiogenic syncope
  * Unstable angina
  * Uncompensated congestive heart failure
  * Poorly controlled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Able to undergo peripheral blood draw

  * No port-a-cath or Hickman catheters
* Planning to reside in the Washington D.C. metro area for at least 1 year after study entry
* Willing to undergo urine testing for cotinine levels and breath testing for carbon monoxide monitoring
* No significant physical or psychological disability that would preclude study participation
* No known allergy to bupropion
* Baseline urine drug screen negative

  * Prescribed pain medication allowed
* None of the following predisposing factors that may increase the risk of seizures with bupropion use:

  * History of seizures
  * Alcohol use > 4 oz/day
  * History of closed head injury
  * History of an eating disorder
  * CNS infection
* No poorly controlled diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 years since prior alcohol abuse or substance abuse therapy (except for tobacco use or dependence)
* More than 14 days since prior monoamine oxidase (MAO) inhibitor
* No concurrent MAO inhibitor
* No concurrent bupropion (Wellbutrin® or Wellbutrin SR®)
* No concurrent alcohol or substance abuse disorder treatment
* No concurrent nicotine replacement therapy
* No concurrent medications that lower seizure threshold (e.g., theophylline or short-acting benzodiazepines)
* No use of tobacco products (more than 1 time per week) other than cigarettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen D. Morgan, PhD, Principal Investigator — NCI - Division of Cancer Control and Population Science; Sandra J. Schaefer, RN, BSN, OCN — National Cancer Institute (NCI)
Locations (1):
- Tobacco Control Research Branch, Rockville, Maryland, United States